CLINICAL TRIAL: NCT02935582
Title: One-year Prospective, Observational Study of the Journey of Patients With Plaque Psoriasis Prescribed Calcipotriol/Betamethasone Aerosol Foam or Other Topical Therapy
Brief Title: PSOREAL - Managing PSOriasis in the REAL World
Acronym: PSOREAL
Status: Completed | Type: Observational
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-ENSTILAR-1285
Record Dates: First submitted 2016-10-14; First posted 2016-10-17 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Psoriasis Vulgaris
Keywords: Topical; Real-world; Local standard of care; Non-interventional; Calcipotriol
MeSH Terms: interventions — calcipotriene

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Enstilar®: Patients for whom a new treatment strategy has been decided which involves start of topical treatment with Enstilar® according to the current local labelling
  Interventions: Drug: Enstilar® aerosol foam
- Other topical: Patients for whom a new treatment strategy has been decided which involves start of topical treatment not including Enstilar®
  Interventions: Drug: Other topical

INTERVENTIONS:
Drug: Enstilar® aerosol foam — Treatment according to local labelling
  Other Names: calcipotriol/betamethasone dipropionate aerosol foam
  Groups: Enstilar®
Drug: Other topical — Treatment according to local practise
  Other Names: Standard topical therapy
  Groups: Other topical

SUMMARY:
Multinational real-life study of current psoriasis treatment strategies, topical treatment patterns and treatment outcomes of these treatments, including the newly introduced calcipotriol/betamethasone dipropionate aerosol foam fixed combination product Enstilar® (calcipotriol/betamethasone dipropionate).

DETAILED DESCRIPTION:
This multinational study aims to describe current treatment patterns and outcomes in the diversity of the real life setting: local differences in access to drugs and current treatment practices, and regional cultural differences, covering adult patients of all backgrounds, sex, socio-economic standing, health background, comorbidity and co-medication. A total of around 400 real-life prescribers in 3-8 countries are expected to participate over the years, with each country contributing data to the study for around 2 years, starting data collection within the first year after local market introduction of Enstilar®.

The real-life prescribing and utilization patterns of topical prescription products approved for treatment of psoriasis vulgaris in the individual participating countries will be mapped and performance of the products in real life will be investigated based primarily on baseline data from investigators and patient reported data contributed by the individual patient for 1 year. Patients are expected to enter data on their electronic device at baseline and at times of treatment changes and other key events, and investigators are expected to contribute data after each contact with the patient.

Patients will be approached for informed consent to participate in the study after their individual treatment plan has been decided. The study aims to include two patients on other topical treatment for every patient planned to receive Enstilar® in order to ensure a sufficient sample of Enstilar® treated patients to capture the diversity of real-life prescription patterns in patients not on Enstilar®, and to allow for sufficiently powered comparisons between Enstilar® and other real-world treatment strategies. A systematic approach will be used to select eligible patients to be approached for study participation in order to minimize selection bias and control seasonal variations.

ELIGIBILITY:
Inclusion Criteria:

* Adult age
* Psoriasis vulgaris
* Plaques on the body (trunk and/or extremities) of at least mild severity at time of inclusion
* Decision to prescribe a topical psoriasis treatment for body use where the prescription is NOT a routine renewal of the prescription of an ongoing therapy
* Signed and dated informed consent
* Willingness and ability to enter personal disease and treatment information onto a secure webpage during the one year individual study period, using their existing access to a PC or electronic device and a personal access code.

Exclusion Criteria:

* Participation in the active treatment phase of a clinical trial
* Previous enrollment in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients starting treatment with Enstilar® or other topical treatment of body and/or extremities in one of the countries participating in the study. Patients receiving a prescription renewal for an ongoing topical treatment are not eligible. Patients undergoing systemic treatment can be included as well, provided they receive a prescription for concomitant use of topical treatment on body and/or extremities and this is not a prescription renewal. The minimum age may vary slightly, as in some countries adult age differ from 18 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 1214 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
PaGA | 4 weeks
  Patient reported Global Assessment
Itch | 1 week
  Itch dimension of Psoriasis Symptom Inventory (PSI) questionnaire
Switch | 1 year
  Time to switch of topical treatment strategy
Flare-up | 1 year
  Time to first flare-up after initial treatment completion

CONTACTS AND LOCATIONS:
Overall Officials: Kreesten M Madsen, MD, PhD, Study Director — LEO Pharma
Locations (3):
- Dr. Chih-Ho Hong Medical Inc., Surrey, British Columbia, Canada
- Psoriasis association in Stockholm region, Stockholm, Sweden
- Layton Medical Centre, Blackpool, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: No